CLINICAL TRIAL: NCT01333046
Title: Administration of Tumor-Associated Antigen (TAA)-Specific Cytotoxic T-Lymphocytes to Patients With Active or Relapsed Hodgkin or Non-Hodgkin Lymphoma
Brief Title: Administration of TAA-Specific CTLs; Hodgkin or Non-Hodgkin Lymphoma; TACTAL
Acronym: TACTAL
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, George Carrum, Associate Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-27471-TACTAL; TACTAL (Other: Baylor College of Medicine); 2P50CA126752-11 (NIH); NCT01556269 (obsolete NCT alias)
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Hodgkin Lymphoma; Non-Hodgkin Lymphoma; Hodgkin Disease
Keywords: Hodgkin Lymphoma; Non-Hodgkin Lymphoma; CTL
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Antigen-Escalation Stage (Experimental): The first stage will be an "antigen-escalation" stage using a fixed total dose of cells (5 x 10^6 cells/m^2 x 2) to evaluate the safety of the T cells primed against PRAME pepmix, and then SSX pepmix, and then MAGE A4 pepmix, and then NY-ESO pepmix, and then SURVIVIN pepmix.
  Interventions: Biological: Antigen-Escalation Stage
- Dose-Escalation Study Stage (Experimental): In the dose escalation stage, three dose levels will be studied. Patients in the dose escalation portion of the study will be entered and stratified separately to the following two groups:
  Group A: Patients receiving CTLs as therapy for Hodgkin's or non-Hodgkin's lymphoma.
  Group B: Patients receiving CTLs as adjunctive therapy following autologous or syngeneic transplant.
  Interventions: Biological: Dose-Escalation Stage
- azacytidine and multiTAA T cells Stage (Experimental): This phase will administer aza intravenously at a dose of 75 mg/m2 after premedication with an anti-emetic such as ondansetron po or IV (up to a maximum dose of 16 mg ondansetron or equivalent). This phase will determine whether infusion of TAA-specific T cells (at dose level 2 - 1x10^7) targeting multiple tumor antigens in combination with azacytidine is safe, and whether CTL infusions (with or without azacytidine) increase the spectrum of epitopes/antigens targeted by endogenous T cells (epitope spreading).
  Interventions: Biological: azacytidine and multiTAA T cells Stage
- Pediatric multiTAA T cells Stage (Experimental): This phase will give patients < 18 years old two infusions (on Day 0 and Day 14) of multi-TAA specific T cells at a fixed dose of 1x10^7 cells/m2. This phase will test the safety and efficacy of multiTAA-specific T cells in pediatric patients with active HL/NHL.
  Interventions: Biological: Pediatric multiTAA T cells Stage

INTERVENTIONS:
Biological: Antigen-Escalation Stage — Antigen-Escalation Stage
  Each patient will receive 2 injections at the same dose (5 x 10^6 cells/m2), 28 days apart, according to the following schedules:
  Schedule One:
  * Day 0: PRAME-specific T cells
  * Day 28: PRAME- and SSX-specific T cells
  Schedule Two:
  * Day 0: PRAME- and SSX-specific T cells
  * Day 28: PRAME/SSX/MAGE-specific T cells
  Schedule Three:
  * Day 0: PRAME/SSX/MAGE-specific T cells
  * Day 28: PRAME/SSX/MAGE/NY-ESO specific T cells
  Schedule Four:
  * Day 0: PRAME/SSX/MAGE/NY-ESO specific T cells
  * Day 28: PRAME/SSX/MAGE/NY-ESO/Survivin-specific T cells
  Other Names: T cell injection; Tumor-specific CTL lines
  Arms: Antigen-Escalation Stage
Biological: Dose-Escalation Stage — Dose-Escalation Stage
  Three different dosing schedules will be evaluated. Each patient will receive 2 injections at the same dose, 14 days apart, according to the following dosing schedules:
  DL1: Day 0 and Day 14: 5 x 10^6 cells/m^2
  DL2: Day 0 and Day 14: 1 x 10^7 cells/m^2
  DL3: Day 0 and Day 14: 2 x 10^7 cells/m^2
  Other Names: TAA-CTL infusion
  Arms: Dose-Escalation Study Stage
Biological: azacytidine and multiTAA T cells Stage — Up to 15 patients will be treated with 3 cycles of aza at a dose of 75 mg/m2 I.V. administered for 5 days/cycle followed, within 28 days of the last aza dose, by two infusions (on Day 0 and Day 14) of multi-TAA specific CTLs at a fixed dose of 1x10^7 cells/m2. If drug-related myelosuppression occurs aza dosing will be modified, according to the following:
  1. ANC >1,000 or Platelets >50,000 (or any other grade I AE attributable to aza)
     Adjustment: None
  2. ANC 500-1000 or Platelets 25,000-50,000 (or any other grade II-III AE attributable to aza)
     Adjustment: 50% dose reduction
  3. ANC <500 or any episode of febrile neutropenia or platelets <25,000 or any episode of bleeding attributed to thrombocytopenia (or any other grade IV or higher AE attributable to aza)
  Adjustment: Discontinue drug, can proceed with CTL infusion if eligible within 28 days of last aza infusion
  Arms: azacytidine and multiTAA T cells Stage
Biological: Pediatric multiTAA T cells Stage — Patients < 18 years old will receive two infusions (on Day 0 and Day 14) of multi-TAA specific T cells at a fixed dose of 1x10^7 cells/m2. We will enroll and infuse at least 5 adolescents on the pediatric arm before opening to all patients.
  Arms: Pediatric multiTAA T cells Stage

SUMMARY:
Patients have a type of lymph gland disease called Hodgkin or non-Hodgkin lymphoma which has come back, or may come back, or has not gone away after treatment, including the standard treatment known for these diseases. This a research study using special immune system cells called tumor associated antigen (TAA)-specific cytotoxic T lymphocytes, a new experimental therapy.

This sort of therapy has been used previously to treat Hodgkin or non-Hodgkin lymphomas that show proof of infection with Epstein-Barr virus (EBV), the virus that causes infectious mononucleosis ("mono" or the "kissing disease"). EBV is found in cancer cells of up to half of all patients with Hodgkin's and non-Hodgkin lymphoma. This suggests that it may play a role in causing lymphoma. The cancer cells infected by EBV are able to hide from the body's immune system and escape being killed. Investigators tested whether special white blood cells, called T cells, that were trained to kill EBV-infected cells could affect these tumors, and in many patients it was found that giving these trained T cells caused a complete or partial response.

However, many patients do not have EBV in their lymphoma cells; therefore investigators now want to test whether it is possible to direct these special T cells against other types of proteins on the tumor cell surface with similar promising results. The proteins that will be targeted in this study are called tumor associated antigens (TAAs) - these are cell proteins that are specific to the cancer cell, so they either do not show or show up in low quantities on normal human cells.

In this study, we will target five TAAs which commonly show on lymphoma, called: NY-ESO-1, MAGEA4, PRAME, Survivin and SSX. This will be done by using special types of T cells called cytotoxic T lymphocytes (CTLs) generated in the lab.

In addition, some adult patients will receive a drug called azacytidine before giving the T cells. We hope that the combination helps the T cells work better.

DETAILED DESCRIPTION:
The patient will give blood to make TAA-specific cytotoxic T cells in the lab. These cells will be grown and frozen. If the TAA-specific cytotoxic T cells can be made, the time from collection of the blood to manufacture of T cells for administration to the patient is about 1 to 2 months.

There are 4 stages of this study: an antigen-escalation phase, a dose-escalation stage, aza stage and pediatric patients stage.

The antigen-escalation phase will be first. Patients will receive TAA-specific T cells targeting first 1 and then 2 TAAs. Once this schedule proves safe, the next group of patients will receive TAA-specific T cells targeting first 2 and then 3 TAAs. This process will continue until all 4 levels are studied. This means that the final cohort of patients will receive TAA-specific T cells targeting first 4 and then 5 TAAs. If the side-effects are too severe, the number of TAAs being targeted will be lowered or the T cell injections will be stopped. Each patient will receive 2 infusions at the same dose 28 days apart

After the antigen-escalation phase, the dose-escalation phase will begin. Patients will be started on the lowest dose (1 of 3 different levels) of T cells. Once that dose schedule proves safe, the next group of patients will be started at a higher dose. This process will continue until all 3 dose levels are studied. If the side-effects are too severe, the dose will be lowered or the T cell injections will be stopped. Each patient will receive 2 infusions at the same dose 14 days apart

After the dose escalation stage, adult patients will be enrolled on the aza stage where they will receive the drug aza followed by two infusions of T cells on dose level 2. Patients will be given 3 cycles of aza (administered daily through a vein for 5 days, every 28 days) followed by 2 doses of multiTAA-specific T cells administered 14 days apart. Before the patient is given the aza they will be given a drug to help prevent nausea and vomiting.

On the pediatric stage, pediatric patients will receive 2 infusions of T cells on dose level 2. The T cells will be given 14 days apart.

The cells will be injected by IV over 10 minutes. The patients may be pre-treated with acetaminophen (Tylenol) and diphenhydramine (Benadryl). Acetaminophen (Tylenol) and diphenhydramine (Benadryl) are given to prevent a possible allergic reaction to the T cell administration. If after the second infusion there is a reduction in the size of the patient's lymphoma on CT or MRI scan as assessed by a radiologist, the patient can receive up to six (6) additional doses of the T cells at monthly intervals if they wish. All of the treatments will be given by the Center for Cell and Gene Therapy at Houston Methodist Hospital or Texas Children's Hospital.

In between the first and second T cell infusions and for 6 weeks after the last infusion, the patient should not receive any other anti-cancer treatments such as radiation therapy or chemotherapy. If the patient does receive any other therapies in-between the first and second infusion of T cells, they will be taken off treatment and will not be able to receive the second infusion of T cells.

MEDICAL TESTS BEFORE TREATMENT

* Physical exam.
* Blood tests to measure blood cells, kidney and liver function.
* Measurements of your tumor by routine imaging studies. We will use the imaging study that was used before to follow your tumor: CT, MRI, or PET.
* Pregnancy test if you are a female who can have children.

MEDICAL TESTS AFTER TREATMENT

- Imaging study 6 weeks after the 2nd TAA-CTL infusion.

To learn more about the way the T cells are working in the patient's body, an extra 20-40 mL (4-8 teaspoons) of blood will be taken before each cycle of aza (if applicable), 2 weeks after each cycle of aza (if applicable), before each T-cell infusion, and at Weeks 1, 2, 4 and 6. One additional blood sample might be drawn 3 to 4 days post the T-cell infusion; this is optional. Afterwards, blood will be collected at 3, 6, 9 and 12 months after the last infusion. The blood may be drawn from a central line at the time of the patient's regular blood tests. Investigators will use this blood to see how long the T cells last,and to look at the immune response to the patient's cancer.

Study Duration: Patients will be on active study participation for approximately one year. Patients who receive additional doses of the T cells as described above will be actively followed until 1 year after their last dose of T cells. Investigators will then remain in contact with patients once a year for up to 4 additional years (total of 5 years follow-up) in order to evaluate disease response long-term.

ELIGIBILITY:
Inclusion Criteria:

PROCUREMENT:

1. Any patient regardless of sex, with a diagnosis of Hodgkin or non-Hodgkin lymphoma.
2. Life expectancy of 6 weeks or greater.
3. Hgb greater than or equal to 7.0
4. Patient and,or parent,guardian able to give informed consent.

TREATMENT:

1. Any patient regardless of sex, with a diagnosis of Hodgkin or non-Hodgkin lymphoma:

   Group A: Patients greater than or equal to 18 years old
   * with active disease:

     * in second or subsequent relapse.
     * in first relapse for indolent lymphoma after first-line therapy for relapse.
     * or first relapse if immunosuppressive chemotherapy contraindicated.
     * primary refractory disease or if persistent disease after first-line therapy of relapse.
   * or multiply relapsed patients in remission who are at a high risk of relapse.
   * or the lymphoma is a second malignancy e.g. a Richters transformation of CLL after failing front line therapy.

   OR

   Group B: Patients greater than or equal to 18 years old after autologous or syngeneic SCT (as adjuvant therapy).

   OR

   Group C: azacytidine plus multiTAA-T cells Patients greater than or equal to 18 years old
   * with active disease in:

     * second or subsequent relapse
     * first relapse for indolent lymphoma after first line therapy for relapse
     * first relapse if immunosuppressive chemotherapy contraindicated
   * with primary refractory disease or persistent disease after first line therapy of relapse
   * or lymphoma as a second malignancy e.g. a Richters transformation of CLL after failing front line therapy

   OR

   GROUP D: Patients less than 18 yrs old
   * with active disease in:

     * second or subsequent relapse
     * first relapse for indolent lymphoma after first line therapy for relapse
     * first relapse if immunosuppressive chemotherapy contraindicated
   * with primary refractory disease or persistent disease after first line therapy of relapse
   * with lymphoma as a second malignancy e.g. a Richters transformation of CLL after failing front line therapy
2. Life expectancy of 6 weeks or greater.
3. Pulse oximetry of more than 95 percent on room air in patients who previously received radiation therapy.
4. Karnofsky,Lansky score of 50 or greater.
5. Creatinine 2X or less of upper limit of normal for age.
6. Patients should have been off other investigational therapy for one month prior to entry in this study.
7. Patients should have been off conventional therapy for at least 1 week prior to entry in this study, including rituximab.
8. Patient and,or parent,guardian able to give informed consent.
9. Due to unknown effects of this therapy on a fetus, pregnant women are excluded from this research. The male partner should use a condom. Females of child-bearing potential should use of at least two forms of contraception unless female has had a hysterectomy or tubal ligation.
10. Bilirubin 2X or less of upper limit of normal, AST 3X or less than the upper limit of normal, and Hgb greater than or equal to 7.0

    GROUP C (aza) Only:
11. Platelets greater than 25,000

Exclusion Criteria:

PROCUREMENT:

1. Patients with severe intercurrent infection.
2. Patients with active HIV infection at time of procurement (can be pending at the time of blood draw).
3. Patients receiving systemic corticosteroids.

TREATMENT:

1. Patients with severe intercurrent infection.
2. Patients receiving systemic corticosteroids.
3. Pregnant breastfeeding.
4. Active viral infection with HIV or hepatitis type B or C. "Active" infection defined as infectious disease testing indicating that patient blood is reactive for Hep B, C and/or HIV and confirmed using PCR to measure viral load.

   GROUP C (aza) Only:
5. Abnormal coagulation parameters (PT greater than 15 seconds, PTT greater than 40 seconds, and/or INR greater than 1.5)
6. Significant active cardiac disease within the previous 6 months including:

   1. NYHA class 4 CHF
   2. Unstable angina
   3. Myocardial infarction
7. Known or suspected hypersensitivity to azacitidine or mannitol
8. Patients with advanced malignant hepatic tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-01; Primary Completion 2021-09-27 (Actual); Study Completion 2027-09-27 (Estimated)

PRIMARY OUTCOMES:
Assessment of patients with adverse events | 8 weeks
  To determine the safety of 2 intravenous injections of autologous TAA-specific cytotoxic T lymphocytes (CTLs) in patients with Hodgkin or non-Hodgkin lymphoma.
Number of Patients with treatment related Serious Adverse Events | 8 weeks
  To determine whether infusion of TAA-specific T cells targeting multiple tumor antigens in combination with azacytidine is safe

SECONDARY OUTCOMES:
Obtain information on the expansion, persistence and anti-tumor effects of the adoptively-transferred TAA-specific CTLs | 1 year
  Information on the expansion, persistence and anti-tumor effects of the adoptively transferred tumor-specific CTLs will be analyzed for the immunological parameters based on multimer analysis, intracellular cytokine staining and ELIspot assays to assess the frequency of cells secreting γ-IFN using the descriptive statistics such as mean, median, standard deviation at each timepoint.
Assessment of increasing the spectrum of epitopes/antigens | 1 year
  To determine whether CTL infusions increase the spectrum of epitopes/antigens targeted by endogenous T cells (epitope spreading).

CONTACTS AND LOCATIONS:
Overall Officials: Geoge Carrum, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Vasileiou S, Lulla PD, Tzannou I, Watanabe A, Kuvalekar M, Callejas WL, Bilgi M, Wang T, Wu MJ, Kamble R, Ramos CA, Rouce RH, Zeng Z, Gee AP, Grilley BJ, Vera JF, Bollard CM, Brenner MK, Heslop HE, Rooney CM, Leen AM, Carrum G. T-Cell Therapy for Lymphoma Using Nonengineered Multiantigen-Targeted T Cells Is Safe and Produces Durable Clinical Effects. J Clin Oncol. 2021 May 1;39(13):1415-1425. doi: 10.1200/JCO.20.02224. Epub 2021 Jan 28. PMID 33507803

DOCUMENTS (1):
  • Informed Consent Form (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT01333046/ICF_000.pdf